CLINICAL TRIAL: NCT00200993
Title: Peripheral Effects of Exercise on Cardiovascular Health (STRRIDE I)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 268
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity; Hyperlipidemia; Insulin Resistance; Metabolic Syndrome X
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity; Hyperlipidemias; Insulin Resistance; Metabolic Syndrome | interventions — Exercise

INTERVENTIONS:
Behavioral: physical activity

SUMMARY:
To investigate the separate effects of the amount of exercise and exercise intensity on cardiovascular risk factors in overweight men and women with mild to moderate dyslipidemia.

DETAILED DESCRIPTION:
BACKGROUND:

Substantial evidence supports a favorable relationships between cardiovascular fitness, physical activity and cardiovascular health. In particular, it is well established that increased levels of physical activity result in favorable improvements in lipid and carbohydrate metabolism. There is also evidence that increased physical activity and cardiovascular fitness have beneficial effects on cardiovascular health independent of the effects on specific cardiovascular risk factors. One hypothesis proposes that the beneficial effects of regular exercise in humans is mediated through peripheral mechanisms, in particular through the chronic adaptations in skeletal muscle to habitual exercise. The exercise exposures required to achieve health benefits in humans are poorly defined and the mechanisms through which these beneficial adaptations occur are poorly understood. The study will investigate the peripheral biological mechanisms through which chronic physical activity alters carbohydrate metabolism and lipid metabolism, resulting in improvements in these parameters of cardiovascular health and fitness in humans.

DESIGN NARRATIVE:

In this clinical trial, Studies of a Targeted Risk Reduction Intervention through Defined Exercise (STRRIDE I), subjects were randomly assigned to one of three graded exercise training regimens or a sedentary control group and asked to train, after an initial ramp period of up to two months, for six months at a given exercise intensity and dose. Parameters reflecting changes in carbohydrate and lipid metabolism were studied at an integrative physiologic level and with measurable biological endpoints in peripheral skeletal muscle (e.g., capillary surface area). It was proposed that the elucidation of the peripheral mechanisms mediating the favorable responses in carbohydrate and lipid metabolism to chronic physical activity would lead to better understanding of the health benefits conferred by physical activity and cardiovascular fitness in humans and point the way toward better exercise recommendations for clients with significant cardiovascular risk factors. The purpose of this study was to investigate the peripheral biological mechanisms through which chronic physical activity altered carbohydrate metabolism and lipid metabolism, resulting in improvements in these parameters of cardiovascular health and fitness in humans. The driving hypothesis was that health benefits derived from habitual exercise were primarily mediated through adaptations occurring in skeletal muscle, probably related to alterations in exposed capillary surface area in skeletal muscle induced by exercise training. The investigators used graded exercise regimens in moderately obese human subjects with mild to moderate lipid metabolic abnormalities to investigate whether induced alterations in skeletal muscle fiber type, metabolic capacity and capillary surface area accounted for favorable alterations in insulin sensitivity and glucose metabolism, lipoprotein levels and lipid metabolism.

ELIGIBILITY:
Inclusion criteria: age 40 to 65 years, sedentary (exercise less than two times per week), overweight or mildly obese (BMI 25 to 35 kg/m2) with mild to moderate lipid abnormalities (either LDL cholesterol 130 to 190 mg/dl; or HDL cholesterol < 40 mg/dl for men, or 5 < 45 mg/dl for women). Women were postmenopausal.

Exclusion criteria: diabetes; hypertension; other metabolic or musculoskeletal diseases; current use of or intent to diet; use of confounding medications; overt presence of coronary heart disease; or unwillingness to be randomized to any group.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Kraus — Duke University

REFERENCES:
- [Background] Johnson JL, Slentz CA, Duscha BD, Samsa GP, McCartney JS, Houmard JA, Kraus WE. Gender and racial differences in lipoprotein subclass distributions: the STRRIDE study. Atherosclerosis. 2004 Oct;176(2):371-7. doi: 10.1016/j.atherosclerosis.2004.05.018. PMID 15380461
- [Background] Hittel DS, Kraus WE, Tanner CJ, Houmard JA, Hoffman EP. Exercise training increases electron and substrate shuttling proteins in muscle of overweight men and women with the metabolic syndrome. J Appl Physiol (1985). 2005 Jan;98(1):168-79. doi: 10.1152/japplphysiol.00331.2004. Epub 2004 Sep 3. PMID 15347626
- [Background] Slentz CA, Duscha BD, Johnson JL, Ketchum K, Aiken LB, Samsa GP, Houmard JA, Bales CW, Kraus WE. Effects of the amount of exercise on body weight, body composition, and measures of central obesity: STRRIDE--a randomized controlled study. Arch Intern Med. 2004 Jan 12;164(1):31-9. doi: 10.1001/archinte.164.1.31. PMID 14718319
- [Background] Houmard JA, Tanner CJ, Slentz CA, Duscha BD, McCartney JS, Kraus WE. Effect of the volume and intensity of exercise training on insulin sensitivity. J Appl Physiol (1985). 2004 Jan;96(1):101-6. doi: 10.1152/japplphysiol.00707.2003. Epub 2003 Sep 12. PMID 12972442
- [Background] Hittel DS, Kraus WE, Hoffman EP. Skeletal muscle dictates the fibrinolytic state after exercise training in overweight men with characteristics of metabolic syndrome. J Physiol. 2003 Apr 15;548(Pt 2):401-10. doi: 10.1113/jphysiol.2002.036616. Epub 2003 Feb 28. PMID 12611918
- [Background] Kraus WE, Houmard JA, Duscha BD, Knetzger KJ, Wharton MB, McCartney JS, Bales CW, Henes S, Samsa GP, Otvos JD, Kulkarni KR, Slentz CA. Effects of the amount and intensity of exercise on plasma lipoproteins. N Engl J Med. 2002 Nov 7;347(19):1483-92. doi: 10.1056/NEJMoa020194. PMID 12421890
- [Background] Kraus WE, Torgan CE, Duscha BD, Norris J, Brown SA, Cobb FR, Bales CW, Annex BH, Samsa GP, Houmard JA, Slentz CA. Studies of a targeted risk reduction intervention through defined exercise (STRRIDE). Med Sci Sports Exerc. 2001 Oct;33(10):1774-84. doi: 10.1097/00005768-200110000-00025. PMID 11581566
- [Background] Slentz CA, Aiken LB, Houmard JA, Bales CW, Johnson JL, Tanner CJ, Duscha BD, Kraus WE. Inactivity, exercise, and visceral fat. STRRIDE: a randomized, controlled study of exercise intensity and amount. J Appl Physiol (1985). 2005 Oct;99(4):1613-8. doi: 10.1152/japplphysiol.00124.2005. Epub 2005 Jul 7. PMID 16002776
- [Background] Duscha BD, Slentz CA, Johnson JL, Houmard JA, Bensimhon DR, Knetzger KJ, Kraus WE. Effects of exercise training amount and intensity on peak oxygen consumption in middle-age men and women at risk for cardiovascular disease. Chest. 2005 Oct;128(4):2788-93. doi: 10.1378/chest.128.4.2788. PMID 16236956
- [Background] Hulver MW, Zheng D, Tanner CJ, Houmard JA, Kraus WE, Slentz CA, Sinha MK, Pories WJ, MacDonald KG, Dohm GL. Adiponectin is not altered with exercise training despite enhanced insulin action. Am J Physiol Endocrinol Metab. 2002 Oct;283(4):E861-5. doi: 10.1152/ajpendo.00150.2002. PMID 12217905
- [Derived] Huffman KM, Koves TR, Hubal MJ, Abouassi H, Beri N, Bateman LA, Stevens RD, Ilkayeva OR, Hoffman EP, Muoio DM, Kraus WE. Metabolite signatures of exercise training in human skeletal muscle relate to mitochondrial remodelling and cardiometabolic fitness. Diabetologia. 2014 Nov;57(11):2282-95. doi: 10.1007/s00125-014-3343-4. Epub 2014 Aug 5. PMID 25091629
- [Derived] Slentz CA, Tanner CJ, Bateman LA, Durheim MT, Huffman KM, Houmard JA, Kraus WE. Effects of exercise training intensity on pancreatic beta-cell function. Diabetes Care. 2009 Oct;32(10):1807-11. doi: 10.2337/dc09-0032. Epub 2009 Jul 10. PMID 19592624